CLINICAL TRIAL: NCT05922540
Title: a Prospective, Multicenter Cohort Study of Ischemic Cerebrovascular Disease
Brief Title: a Cohort Study of Ischemic Cerebrovascular Disease
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 202304068
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Ischaemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- those with favorable prognosis
  Interventions: Other: Intravenous thrombolysis
- those with unfavorable prognosis
  Interventions: Other: Intravenous thrombolysis

INTERVENTIONS:
Other: Intravenous thrombolysis — Intravenous thrombolysis with alteplase within the time window of stroke onset in stroke patients

SUMMARY:
This study aims to establish a multicenter, large-scale, prospective cohort of patients with ischemic stroke. Various biological samples such as blood, feces, and urine are collected to identify biomarkers associated with ischemic stroke. By integrating demographic information, clinical indicators, imaging parameters, and biomarker parameters, the study aims to develop risk assessment, early warning, and prognosis prediction models. Additionally, the study aims to identify key genes and explore relevant signaling pathways related to ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of ischemic stroke.
2. Age ≥ 18 years.
3. Signed informed consent form.

Exclusion Criteria:

1. Patients with moderate to severe mental disorders or dementia who cannot cooperate to complete the informed consent and follow-up procedures.
2. Patients with neurological functional impairment caused by conditions such as migraine aura, epilepsy, or other non-ischemic strokes.
3. Agitated patients who cannot cooperate with imaging examinations.
4. Pregnant or lactating patients, as well as those planning to become pregnant within 90 days.
5. Patients with concurrent malignant tumors or severe systemic diseases with an expected survival period of less than 90 days.
6. Patients who have participated in other clinical studies within 30 days prior to enrollment or are currently participating in other interventional clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Continuously enroll hospitalized patients who meet the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Cerebrovascular events | 3 months of onset in patients
  Cerebrovascular events, including ischemic stroke, transient ischemic attack, cerebral hemorrhage, subarachnoid hemorrhage
mRS scores | 3 months of onset in patients
  Assessing patients' neurological functional impairment status using the mRS score

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Central South University, Hunan, China

IPD SHARING:
Plan to Share IPD: No
Privacy and Confidentiality: Sharing IPD may raise concerns regarding the privacy and confidentiality of the participants. Protecting the personal information and identities of the participants is a priority, and sharing IPD may involve potential risks in this regard.